CLINICAL TRIAL: NCT06111456
Title: Acceptability of Expanded Newborn Screening to Parents in France With or Without Genetics in the First Line
Acronym: SeDeN-p3
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: OLIVIER-FAIVRE 2021-2
Record Dates: First submitted 2023-10-18; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Expanded Newborn Screening; Parental Acceptability
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Population 1Q: Parents or co-parents of a newborn child.
  Interventions: Other: Questionnaire; Other: Interview
- Population 2: Parents or co-parents whose youngest child is 1 week to 3 years old.
  Interventions: Other: Questionnaire
- Population 3: Parents or co-parents whose child had a suspicious newborn screening result that was confirmed at the diagnosis phase (except hearing).
  Interventions: Other: Interview
- Population 4: Parents or co-parents whose child was diagnosed later based on clinical signs for diseases not included in the list of diseases screening in French newborn screening, but included in the list of diseases screened in newborn screening in other countries.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Questionnaire — Online self-administered questionnaire to quantitatively mesure parental knowledge and expectations on current and expanded newborn screeing and parental acceptability of expanded newborn screening using genetic.
  Groups: Population 1Q; Population 2
Other: Interview — Semi-structured interview to explore parental representations on the extension of newborn screening and - if concerned - to retrace the screening/diagnosis/care management pathway
  Groups: Population 1Q; Population 3; Population 4

SUMMARY:
The recent modifications of the French bioethics law, the therapeutic progress and the massive development of advanced genetic techniques (such Next-Generation Sequencing (NGS)) with a rapid decrease in costs imply to question the extension of Newborn Screening (NBS) to new actionable pathologies and the acceptable and relevant methods for its possible expansion. International studies are beginning to determine the potential place of NGS in NBS. In this perspective, the SeDeN project aims to fully assess the social acceptability of these issues by measuring the diversity and consistency of expectations of French health professionals, parents and public policy makers.

The SeDeN-p3 Study focuses on the opinions of parents. It aims to analyze the perception of parents in different situations: birth, early childhood, child screened in the framework of the national neonatal screening program, etc. The objective of this part is to study the understanding and expectations of parents in France regarding the extension of newborn screening as well as their preferences regarding its conditions (information, types of pathologies, screening methods, etc.).

ELIGIBILITY:
Inclusion Criteria:

All populations combined:

* Be a parent or co-parent
* Age of parent:

  * woman between 18 and 50 years
  * man between 18 and 60 years
* Live in metropolitan France
* Have received information about the SeDeN-p3 Study
* Understand the purpose of the SeDeN-p3 Study

Self-administered questionnaire:

* Be able to read and answer a self-administered questionnaire in French

  * Population 1Q:
* Have a child less than a week old
* Have just giver birth in 1 of the partner maternity hospitals during the survey period

  * Population 2:
* Parent or co-parent whose youngest child is between 1 week and 3 years old
* Be part of the panel of the selected survey-sample firm

Semi-structured interviews

* Can converse fluently in French
* Accept to conduct a recorded interview

  * Population 1E (sub-population of Population 1Q)
* Have completed the entire questionnaire

  * Population 3
* Have a child under 5 years old (inclusive) with 1 of the following diseases :

  * Phenylketonuria
  * Congenital hypothyroidism
  * Congenital adrenal hyperplasia
  * Cystic fibrosis
  * Sickle cell disease
  * hearing loss
  * MCAD deficiency
  * glutaric aciduria type -1
  * isovaleric academia
  * LCHAD deficiency
  * carnitine deficiency
  * homocystinuria
  * leukinosis
  * tyrosinemia type 1

    * Population 4
* Have a child under 17 years old (inclusive), with 1 of following diseases:

  * Citrullinemia type I
  * Ornithine Transcarbamylase Deficiency
  * Methylmalonic acidaemia
  * Very long-chain acyl-CoA dehydrogenase deficiency
  * Carnitine palmitoyl transferase 1 deficiency
  * Carnitine palmitoyl transferase 2 deficiency
  * Glutaric acidaemia type II
  * Galactosaemia
  * Biotinidase deficiency
  * Pompe Disease
  * Mucopolysaccharidosis Type 1
  * Glucose-6-phophate dehydrogenase deficiency
  * X-linked Adrenoleukodystrophy
  * Spinal muscular atrophy linked to SMN1
  * S, beta-thalassemia

Exclusion Criteria:

* Have a newborn child die during the recruitment period
* Not speak and/or understand French
* Refuse to participate in the SeDeN-p3 Study
* Be under judicial protection (tutelle, curatelle, habilitation familiale et sauvegarde de justice)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Parents or co-parents in France with a sick child or not
Sampling Method: Non-Probability Sample
Enrollment: 1585 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Mixed matrix of parental acceptability dimensions of expanded newborn screening (Mixed-data matrix) | November 2023
  Mixed method design used to measure parental acceptability composed of quantitative and qualitative data

SECONDARY OUTCOMES:
Parental acceptability scores for expanded newborn screening (Theorical Framework of Acceptability scores in self-administered questionnaire to measure parental acceptability) | November 2023
Typology of parental acceptability scores for expanded newborn screening (Classification) | November 2023
Measure of importance given to different modalities of information about newborn screening (by whom, when, how, etc.) (Multiple Choice Questions) | November 2023
Parent opinion on newborn screening for Spinal Muscular Atrophy, Duchenne muscular dystrophy, BRCA-related breast and ovarian cancer predisposition syndrome and congenital long QT | November 2023
  (5-point Likert scale for agreement and thematic content analysis of the free comment areas)
Parent's views on the use of genetic testing in expanded newborn screening (Likert scales) | November 2023
Description of acceptability of expanded newborn screening to parents of a sick child (Thematic content analysis) | April 2024

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hopital Antoine Beclere - Aphp, Clamart
  - Chu Dijon Bourgogne, Dijon
  - Hôpital Necker - Enfants Malades, Paris
  - Groupe Hospitalier de La Haute-Saône, Vesoul